CLINICAL TRIAL: NCT06117904
Title: Assessing the Effects and Safety of MEBO as Add on Therapy for the Prevention of Radiotherapy-Induced Mucositis
Brief Title: Adjunctive Treatments for the Prevention of Radiotherapy-Induced Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelfattah Elsayed, Lecturer of clinical pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BeniSuefUU
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Radiotherapy Side Effect; Mucositis
MeSH Terms: conditions — Radiation Injuries; Mucositis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEBO ointment + symptomatic therapy (Experimental): This group included twenty-five patients given Mebo ointment in combination with the symptomatic therapy 3 times daily for 7 weeks.
  Interventions: Drug: MEBO ointment; Drug: Symptomatic treatment only
- symptomatic therapy (Active Comparator): This group included twenty-five patients given symptomatic therapy 3 times daily for 7 weeks.
  These therapies included anti-fungal agents (Miconaz oral gel), topical anesthetics and anti-inflammatory drugs (BBC oral spray), topical analgesic gel (Oracure gel), sodium bicarbonate mouthwash (Alkamisr sachets).
  Interventions: Drug: Symptomatic treatment only

INTERVENTIONS:
Drug: MEBO ointment — This group included twenty-five patients given Mebo ointment in combination with the symptomatic therapy 3 times daily for 7 weeks
  Arms: MEBO ointment + symptomatic therapy
Drug: Symptomatic treatment only — This group included twenty-five patients given symptomatic therapy 3 times daily for 7 weeks.
  These therapies included anti-fungal agents (Miconaz oral gel), topical anesthetics and anti-inflammatory drugs (BBC oral spray), topical analgesic gel (Oracure gel), sodium bicarbonate mouthwash (Alkamisr sachets).

SUMMARY:
Radiation therapy (RT) is used in at least 50% of cancer patients and is critical in treating and palliating tumor-related symptoms. Normal tissue radiation toxicity remains an overwhelming obstacle in treating cancer patients with localized tumors.

Mucositis is the inflammation and ulceration of the oral and gastrointestinal mucosa observed with different cancer therapies. Oral mucositis is a common, severe, and debilitating complication of RT occurring several days to weeks after RT initiation.

DETAILED DESCRIPTION:
This study is a single blind randomized controlled clinical trial with a parallel-group design conducted in the clinical oncology department of Beni-Suef University Hospital.

A total of 50 patients with head and neck cancer receiving RT were randomly assigned into either study group:

Group 1 (Intervention group):

This group included twenty-five patients given Mebo ointment in combination with the symptomatic therapy 3 times daily for 7 weeks

Group 2 (Control group):

This group included twenty-five patients given symptomatic therapy 3 times daily for 7 weeks.

These therapies included anti-fungal agents (Miconaz oral gel), topical anesthetics and anti-inflammatory drugs (BBC oral spray), topical analgesic gel (Oracure gel), sodium bicarbonate mouthwash (Alkamisr sachets)

1. Oral mucositis severity was measured by the World Health Organization Toxicity Scale (WHO grading system). Based on the symptomatic (oral pain), and functional clinical features of every patient (ability to drink and eat) as well as the presence of lesions (ulcers, erythema), the measurements were categorized to Grade I: presence of soreness and erythema, Grade II: presence of painful erythema and ulcerations that do not affect the patient solid food intake, Grade Ш: confluent ulceration that affect the solid food intake and require liquid diet, and Grade ΙV: the patient requires parenteral nutrition.
2. Discomfort and pain severity were recorded using the Numeric Rating Scale (NRS), which is categorized to no pain (NRS 0), mild pain (NRS 1-3), moderate pain (NRS 4-7), and unbearable pain (NRS 8-10). Patients were asked to assign a numerical score on the scale verbally to rate their pain intensity, and the number was recorded
3. Dry mouth, Dysphagia was measured by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.

Grade 2 Moderate; minimal, local or noninvasive intervention indicated. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care.

Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (>18 years) with histopathologically confirmed Head and Neck Cancer (HNC), primary tumor in the stages T1, T2, T3, or T4, a regional node of any N status, and distant metastases absent.
2. All patients who were going to receive RT (dose between 60-70 Gy) on the head and neck region as postoperative (adjuvant) or definitive therapy. Either these patients had received chemotherapy prior or in concomitant to radiotherapy.
3. Eastern Cooperative Oncology Group (ECOG) performance score (PS) of 0 to 2 and normal hematologic and biochemical parameters.

Exclusion Criteria:

1. patients undergoing previous radiotherapy
2. uncontrolled systemic or widely disseminated disease
3. having any physical or mental abnormality,
4. pregnant and lactating women
5. presence of a synchronous double primary malignancy or simultaneous participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Oral mucositis Severity | 7 weeks
  Oral mucositis severity was measured by the World Health Organization Toxicity Scale (WHO grading system) Grade 1 Mild; asymptomatic Grade 2 Moderate; minimal, local inflammation Grade 3 Severe or medically significant Grade 4 Life-threatening Grade 5 Death

SECONDARY OUTCOMES:
Dry mouth, Dysphagia score | 7 weeks
  Dry mouth, Dysphagia was measured by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 Grade 1: Symptomatic, able to eat regular diet Grade 2: Symptomatic and altered eating/swallowing Grade 3: Severely altered eating/swallowing; tube feeding, TPN, or hospitalization indicated Grade 4: Life-threatening consequences; urgent intervention indicated Grade 5: Death
Discomfort and pain severity | 7 weeks
  Discomfort and pain severity were recorded using the Numeric Rating Scale (NRS) Grade 1: Mild pain Grade 2: Moderate pain Grade 3: Severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Engy Wahsh, Study Director — 6october University
Locations (1):
- Asmaa Abdelfattah Elsayed, Banī Suwayf, Egypt

REFERENCES:
- [Background] Delaney G, Jacob S, Featherstone C, Barton M. The role of radiotherapy in cancer treatment: estimating optimal utilization from a review of evidence-based clinical guidelines. Cancer. 2005 Sep 15;104(6):1129-37. doi: 10.1002/cncr.21324. PMID 16080176
- [Background] Saadeh CE. Chemotherapy- and radiotherapy-induced oral mucositis: review of preventive strategies and treatment. Pharmacotherapy. 2005 Apr;25(4):540-54. doi: 10.1592/phco.25.4.540.61035. PMID 15977916